CLINICAL TRIAL: NCT00713778
Title: The Impact of Electrocoagulation on Ovarian Reserve After Laparoscopic Exc
Brief Title: The Impact of Electrocoagulation on Ovarian Reserve After Laparoscopic Excision of Ovarian Cyst
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Shandong University (Other)
Responsible Party: Xiayong Wang Ph.D, Shandong Provincial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SPH-CL-030408
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-07

CONDITIONS: Ovarian Cysts
Keywords: Ovarian Cysts; Electrocoagulation; Ovarian Function Tests; Laparoscopy
MeSH Terms: conditions — Ovarian Cysts; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Laparoscopic ovarian cystectomy using bipolar
  Interventions: Procedure: Ovarian cystectomy
- 2 (Experimental): Laparoscopic ovarian cystectomy using ultrasonic scalpel
  Interventions: Procedure: Ovarian cystectomy
- 3 (Active Comparator): Laparotomic ovarian cystectomy using suture
  Interventions: Procedure: Ovarian cystectomy

INTERVENTIONS:
Procedure: Ovarian cystectomy — Laparoscopic ovarian cystectomy using bipolar
  Other Names: laparoscopic ovarian cystectomy using bipolar
  Arms: 1
Procedure: Ovarian cystectomy — Laparoscopic ovarian cystectomy using ultrasonic scalpel electrocoagulation
  Other Names: laparoscopic ovarian cystectomy using ultrasonic scalpel
  Arms: 2
Procedure: Ovarian cystectomy — Laparotomic ovarian cystectomy using suture
  Other Names: Laparotomic ovarian cystectomy using suture
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the impact of electrocoagulation on ovarian reserve after laparoscopic excision of ovarian cyst and the possible mechanisms.

DETAILED DESCRIPTION:
Laparoscopic cystectomy is currently considered the treatment of choice in women with benign ovarian cysts and has gained increasing acceptance among gynecological surgeons(1). However, the safety of this technique in terms of ovarian damage to the operated gonad has recently been questioned. In the present study, with the combined use of serum hormonal evaluation and ultrasound examination, we planned to prospectively investigate the ovarian reserve after the excision of benign ovarian cysts. The damage to ovarian reserve will be evaluated through a 12-months follow-up after the application of bipolar, ultrasonic scalpel electrocoagulation or suture during ovarian cystectomy

ELIGIBILITY:
Inclusion criteria:

* Age 18-40 years
* Uni/bilateral ovarian cyst(s) without clinical and sonographic suspicion of ovarian cancer
* Regular menstrual cycles defined as cycle length between 25 and 35 days in the 6 months before surgery
* Agreement to be enrolled in the study

Exclusion criteria:

* Prior ovarian surgery
* Surgical necessity to perform adnexectomy
* Known endocrine disease
* Post operative pathologic diagnosis was not benign ovarian cyst
* Oral contraceptive use before surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2003-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Serum FSH and E2 assays | 12 months

SECONDARY OUTCOMES:
Transvaginal ultrasound examinations for basal antral follicle number, mean ovarian diameter and peak systolic velocity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: changzhong li, M.D., Study Director — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

REFERENCES:
- [Background] Candiani M, Barbieri M, Bottani B, Bertulessi C, Vignali M, Agnoli B, Somigliana E, Busacca M. Ovarian recovery after laparoscopic enucleation of ovarian cysts: insights from echographic short-term postsurgical follow-up. J Minim Invasive Gynecol. 2005 Sep-Oct;12(5):409-14. doi: 10.1016/j.jmig.2005.06.006. PMID 16213426
- [Background] Ho HY, Lee RK, Hwu YM, Lin MH, Su JT, Tsai YC. Poor response of ovaries with endometrioma previously treated with cystectomy to controlled ovarian hyperstimulation. J Assist Reprod Genet. 2002 Nov;19(11):507-11. doi: 10.1023/a:1020970417778. PMID 12484492
- [Background] Loh FH, Tan AT, Kumar J, Ng SC. Ovarian response after laparoscopic ovarian cystectomy for endometriotic cysts in 132 monitored cycles. Fertil Steril. 1999 Aug;72(2):316-21. doi: 10.1016/s0015-0282(99)00207-1. PMID 10439003
- [Background] Nargund G, Cheng WC, Parsons J. The impact of ovarian cystectomy on ovarian response to stimulation during in-vitro fertilization cycles. Hum Reprod. 1996 Jan;11(1):81-3. doi: 10.1093/oxfordjournals.humrep.a019043. PMID 8671163
- [Background] Somigliana E, Ragni G, Benedetti F, Borroni R, Vegetti W, Crosignani PG. Does laparoscopic excision of endometriotic ovarian cysts significantly affect ovarian reserve? Insights from IVF cycles. Hum Reprod. 2003 Nov;18(11):2450-3. doi: 10.1093/humrep/deg432. PMID 14585900